CLINICAL TRIAL: NCT01272882
Title: Electrical Impedance Tomography (EIT) Monitoring: A Pilot Comparison to Standard of Care Assessments in Adults With Acute Lung Injury (ALI) or Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Electrical Impedance Tomography (EIT) Monitoring in Adults With ALI or ARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CCC#30067; DDD# 600788 (Other: DDD# 600788)
Record Dates: First submitted 2011-01-03; First posted 2011-01-10 (Estimated); Results first posted 2013-01-07 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-04

CONDITIONS: Acute Lung Injury (ALI); ARDS
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adults with ARDS or ALI (Experimental): Adults with PaO2/FiO2 ratio less than 300. Consented patients will be placed on EIT monitor. The only intervention is the addition of Electrical Impedance Tomography monitoring using the Chest belt with 16 electrodes connected to the EIT device. No changes to standard patient care will occur other than collecting EIT monitor data.
  Interventions: Device: Electrical Impedance Tomography monitoring

INTERVENTIONS:
Device: Electrical Impedance Tomography monitoring — Chest belt with 16 electrodes connected to the EIT device

SUMMARY:
Electrical impedance tomography (EIT) monitoring has been researched as a method to determine the spatial impedance distribution in a body cross section, but has yet to become an established clinical tool. EIT monitoring gives a dynamic, breath-to-breath measurement of both global and regional ventilation. Recently, there has been evidence that EIT monitoring has great potential to become a non-invasive bedside tool for assessment of regional lung ventilation without documented hazards. Potential applications include any adult patients in acute respiratory failure. Data collected from this research may contribute to improved patient safety outcomes.

PURPOSE:

The purpose of this pilot study is to examine the feasibility of using the EIT monitor in intensive care unit (ICU) setting on patients with acute respiratory failure and to compare the EIT monitor data to standard of care patient assessments. It is hypothesized that the EIT monitor, when applied to adults in acute respiratory failure, will correlate with conventional standard of care assessments for these patients.

DETAILED DESCRIPTION:
INTRODUCTION:

Electrical impedance tomography (EIT) monitoring has been researched as a method to determine the spatial impedance distribution in a body cross section, but has yet to become an established clinical tool. EIT monitoring gives a dynamic, breath-to-breath measurement of both global and regional ventilation. Recently, there has been evidence that EIT monitoring has great potential to become a non-invasive bedside tool for assessment of regional lung ventilation without documented hazards. Potential applications include any adult patients in acute respiratory failure. Data collected from this research may contribute to improved patient safety outcomes.

PURPOSE:

The purpose of this pilot study is to examine the feasibility of using the EIT monitor in ICU setting on patients with acute respiratory failure and to compare the EIT monitor data to standard of care patient assessments. It is hypothesized that the EIT monitor, when applied to adults in acute respiratory failure, will correlate with conventional standard of care assessments for these patients.

METHOD:

This pilot study design will consist of a prospective, blinded evaluation of the EIT monitor for patients with acute lung injury or acute respiratory distress syndrome.

Once a patient has met the inclusion criteria and has signed informed consent:

1. EIT electrode chest band will be applied by trained respiratory care staff. Application includes elastic chest band with 16 electrodes.
2. EIT electrode chest band is connected to the EIT monitor which will be turned on and will monitor and store EIT data.
3. EIT monitoring will take place for 4 to 6 hours, during day shift (7am to 4pm)
4. Patient's may be monitored on three separate days.

No interventions, tests or modifications to the standard of care will occur to patients for this pilot study of EIT monitoring. Clinicians guiding the care of these patients will be blinded to the EIT data. The EIT chest band will be removed if transport of the patient is necessary or if care is needed in the area of the chest band.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in this study if the following criteria have been met:

1. Males and females > 18 years old (non-pregnant, non-lactating females).
2. Partial pressure of arterial oxygen (PaO2) / Fraction of inspired oxygen (FiO2) ratio < 300 torr.
3. Signed informed consent has been obtained.

Exclusion Criteria:

1. Females who are pregnant or lactating.
2. Patients with skin abrasions or wounds in the chest area.
3. Patients receiving dialysis.
4. Patients with pacemakers or paced EKG rhythms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John S Emberger, BS, Principal Investigator — Christiana Care Health Services; Vinay Maheshwari, MD, Principal Investigator — Christiana Care Health Services; Joel M Brown, BS, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Hospital, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No
IPD data will not be shared

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Intensive care units
Pre-assignment Details: No pre-assignment details to note.
Groups:
- Adults With ARDS or ALI: Adults with PaO2/FiO2 ratio less than 300.
  Electrical Impedance Tomography monitoring : Chest belt with 16 electrodes connected to the EIT device
Period: Overall Study
Arm/Group | Adults With ARDS or ALI
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Adults With ARDS or ALI
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of EIT Monitoring in This Population of ARDS/ALI Patients
Description: Feasibility for the purposes of our study was the ability to apply the device to a diverse population of ARDS/ALI patients and obtain EIT data from the device.
Time Frame: At the start of monitoring once the patient was consented and enrolled.
Measure: Number; unit: Patients successfully monitored with EIT
Arm/Group | Adults With ARDS or ALI
Number analyzed (Participants) | 13
Patients successfully monitored with EIT | 13

ADVERSE EVENTS:
Arm/Group | Adults With ARDS or ALI
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes